CLINICAL TRIAL: NCT03756545
Title: Neurobehavioral Moderators of Post-traumatic Disease Trajectories: Prospective MRI Study of Recent Trauma Survivors
Brief Title: Neurobehavioral Moderators of Post-traumatic Disease Trajectories
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: New York University (Other); Texas A&M University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, michal roll, Prof. Talma Hendler, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0207-14-TLV; R01MH103287 (NIH)
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: PTSD; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research goal is to uncover the neurocognitive moderators of PTSD trajectories, by documenting clinical symptoms, cognitive functioning, and brain structure and function, one-, six- and fourteen months following a traumatic event, in a large population of survivors at initial high risk for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Able to read and comprehend Hebrew
* Arrived in the ER because of one of the following: car accidents, terrorist attacks, work accidents, home accidents, burns, physical assault, large-scale disaster.

Exclusion Criteria:

* Individuals with known claustrophobia
* Individuals with history of substance abuse
* Individuals with current or past psychotic or bipolar I disorder
* Individuals with chronic PTSD at the time of the current trauma
* Individuals on psychotropic medication or recreational drugs in the week that precedes the MRI
* Individuals with hearing problems
* Individuals with head trauma with coma exceeding 30 minutes
* Individuals which can't perform MRI due to safety reasons (e.g. irremovable metals in their body)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult civilians admitted to Tel-Aviv Sourasky Medical Center's Emergency Room (ER), following a potentially traumatic incident. The initial screening will be done via telephone-based structured interviews within 10 days of ER admission, in order to confirm the occurrence of psychologically traumatic event, identify & assess those expressing initial Acute Stress Disorder (ASD) symptoms.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Change in CAPS Total Scores | one-, six- and fourteen months following a traumatic event
  The Clinician-Administered PTSD Scale, used to assess PTSD diagnostic status and symptom severity. CAPS total symptom severity score is calculated by summing severity scores for all PTSD symptoms. We use both CAPS-V (according to DSM-4) and CAPS-5 (according to DSM-5).

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Y Shalev, Prof., Principal Investigator — Department of Psychiatry, NYU Langone Medical Center, New York, NY, United States
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Ben-Zion Z, Spiller TR, Keynan JN, Admon R, Levy I, Liberzon I, Shalev AY, Hendler T, Harpaz-Rotem I. Evaluating the Evidence for Brain-Based Biotypes of Psychiatric Vulnerability in the Acute Aftermath of Trauma. Am J Psychiatry. 2023 Feb 1;180(2):146-154. doi: 10.1176/appi.ajp.20220271. Epub 2023 Jan 11. PMID 36628514
- [Derived] Sheynin S, Wolf L, Ben-Zion Z, Sheynin J, Reznik S, Keynan JN, Admon R, Shalev A, Hendler T, Liberzon I. Deep learning model of fMRI connectivity predicts PTSD symptom trajectories in recent trauma survivors. Neuroimage. 2021 Sep;238:118242. doi: 10.1016/j.neuroimage.2021.118242. Epub 2021 Jun 5. PMID 34098066
- [Derived] Ben-Zion Z, Artzi M, Niry D, Keynan NJ, Zeevi Y, Admon R, Sharon H, Halpern P, Liberzon I, Shalev AY, Hendler T. Neuroanatomical Risk Factors for Posttraumatic Stress Disorder in Recent Trauma Survivors. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Mar;5(3):311-319. doi: 10.1016/j.bpsc.2019.11.003. Epub 2019 Nov 20. PMID 31973980